CLINICAL TRIAL: NCT03453034
Title: To Study the Pharmacokinetic Characteristics of TQ-B233 in the Human Body, Recommend a Reasonable Regimen for Subsequent Research
Brief Title: Tolerance and Pharmacokinetics of TQ-B3233
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TQ-B3233-I-01
Record Dates: First submitted 2017-12-23; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Tumor
Keywords: TQ-B3233; tumor; toleration; pharmacokinetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3233 capsule (Experimental): QD or BID; patients are given the doses according to the protocal, and a cycle is 28 days.
  Interventions: Drug: TQ-B3233

INTERVENTIONS:
Drug: TQ-B3233 — QD or BID in different stage of this research

SUMMARY:
Study of Tolerance and Pharmacokinetics of TQ-B3233 Capsule, phase I,single arm.

DETAILED DESCRIPTION:
The maximum tolerated dose (MTD) of TQ-B3233 [ Time Frame: 48 weeks ] [ Designated as safety issue: Yes ]The highest dose at which no more than 33% of the subjects experience a dose-limiting toxicity (DLT) during treatment.

Pharmacokinetics of TQ-B3233 (in whole blood):In the study of single-dose, full PK profiles will be obtained at H0/H0.5/H1/H2/H3/H5/H8/H10/H12/H24/H48/H72（H means Hour）.In the study of multiple-dose,full PK profiles will be obtained at D0/D1/D2/D8/D15/D22/D28（D means Day）.

ELIGIBILITY:
Inclusion Criteria:

* Patients definitely diagnosed by pathology and/or cytology as BRAF mutation advanced malignant melanoma.
* 18-70 years old, ECOG PS:0-1,Life expectancy of more than 3 months;
* Patients treated with chemotherapy agents or surgery before being enrolled into the study need waiting for 4 weeks, 6 weeks will be needed if agents were nitrocarbamide and mitomycin C;
* Main organs function is normal;
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped;
* Patients should be voluntary and sign the informed consent before taking part in the study;

Exclusion Criteria:

* Patients with Malignant tumors within 5 years, except for non-melanoma skin cancer and in situ cancer;
* Patients who had previously received specific BRAF inhibitors;
* A variety of factors that affect oral medication (such as inability to swallow, gastrointestinal resection, chronic diarrhea, intestinal obstruction, etc.)
* Patients who participated in other anticancer drug clinical trials within 4 weeks ;
* Blood pressure unable to be controlled ideally by one drug(systolic pressure≥150 mmHg，diastolic pressure≥90 mmHg);
* Patients with Grade 1 or higher myocardial ischemia, myocardial infarction or malignant arrhythmias or cardiac insufficiency (including QTc≥480ms) and patients with Grade 3 or higher congestive heart failure (NYHA Classification);
* Patients with non-healing wounds or fractures;
* Patients with brain metastasis, spinal cord compression, cancerous meningitis, CT or MRI examination reminds patients with cerebral or soft meningeal diseases in the screening phase;
* Patients with drug abuse history or unable to get rid of drugs or Patients with mental disorders;
* Coagulation function abnormality: haemorrhagic tendencies (e.g. active digestive tract ulcer), or are receiving thrombolytic or anticoagulant therapy;
* Patients with immunodeficiency, including HIV positive or other acquired, congenital immunodeficiency disease, or organ transplant history;
* Patients with thyroid dysfunction;
* Patients with concomitant diseases which could seriously endanger themselves or those who won't complete the study according to investigators;
* Parents with hepatitis b surface antigen positive or HCV;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose(MTD) | 28 Days
dose-limiting toxicity(DLT) | 28 Days
Peak Plasma Concentration(Cmax) | up to 28 Days
Peak time(Tmax) | up to 28 Days
Half life(t1/2) | up to 28 Days
Area under the plasma concentration versus time curve (AUC) | up to 28 Days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing cancer hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No